CLINICAL TRIAL: NCT05797558
Title: Unilateral Primary Aldosteronism, Mineralocorticoid Antagonists Versus Surgical Treatment - A Randomized Controlled Trial
Brief Title: Unilateral Primary Aldosteronism, Mineralocorticoid Antagonists Versus Surgical Treatment
Acronym: UPA-MEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Karolinska Institutet (Other); Umeå University (Other)
Responsible Party: Principal Investigator, Oskar Ragnarsson, MD, PHD, Associate Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFGBG-978940; DNR 2020-02008 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2023-02-05; First posted 2023-04-04 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Primary Hyperaldosteronism Due to Adrenal Adenoma
Keywords: hyperaldosteronism; primary aldosteronism; lateralized aldosteronism; unilateral aldosteronism; eplerenone; spironolactone; randomized trial; quality of life; PASO outcomes
MeSH Terms: conditions — Hyperaldosteronism | interventions — Surgical Procedures, Operative; Eplerenone; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: Unblinded, prospective, multi-center,randomized, controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgically Treated Primary Aldosteronism (Active Comparator): Standard therapy
  Interventions: Procedure: Unilateral adrenalectomy
- Medically Treated Unilateral Primary Aldosteronism (Active Comparator): Open label eplerenone treatment
  Interventions: Drug: Medical treatment (eplerenone)

INTERVENTIONS:
Procedure: Unilateral adrenalectomy — Minimally invasive surgery is performed via the lateral transperitoneal approach or the posterior retroperitoneal approach, with or without robotic assistance, according to the surgeon's preference.
  Other Names: Surgery
  Arms: Surgically Treated Primary Aldosteronism
Drug: Medical treatment (eplerenone) — The initial dose of eplerenone is 25 mg twice daily. The dose will be increased by 50 mg every fourth week until systolic blood pressure of 140 mmHg and diastolic blood pressure of 90 mmHg or lower has been reached and biochemical control (plasma renin above the middle of the reference range, i.e > ~20 mIU/L) is attained and/or hyperkalemia develops. The maximal dose of eplerenone is 300 mg twice daily.
  Other Names: Mineralocorticoid receptor antagonists
  Arms: Medically Treated Unilateral Primary Aldosteronism

SUMMARY:
This is a prospective randomized controlled trial where quality of life and the effectiveness of treatment will be evaluated in 80 patients with confirmed unilateral primary aldosteronism ,randomly assigned to be either treated surgically with unilateral adrenalectomy or to receive medical treatment with eplerenone.

DETAILED DESCRIPTION:
Background

Primary aldosteronism (PA) is caused by hypersecretion of the adrenal hormone aldosterone and is the most common cause of secondary hypertension . The estimated prevalence of PA is 5-13% in the hypertensive population.

In half of the cases, PA is caused by unilateral hypersecretion of aldosterone, most commonly from an aldosterone producing adenoma. Overproduction from both adrenals is seen in the other half, usually caused by bilateral idiopathic hyperplasia. Unilateral adrenalectomy is considered to be the treatment of choice for unilateral PA and mineralocorticoid receptor antagonists (MRAs, i.e. spironolactone or eplerenone) for bilateral PA . Untreated PA is associated with a greatly increased risk for several comorbidities, especially cardiovascular diseases and renal failure, as well as death.

Studies comparing surgical and medical treatment for PA are scarce. Nevertheless, a recent meta-analysis indicated that cardiovascular outcome is better in surgically than medically treated patients . In addition, quality of life seems to improve more after surgery, and the need for antihypertensive medications, and overall health care consumption,seems to be lower following surgery . However, suboptimal dosing of MRA is common in medically treated patients with PA, which makes a fair comparison between surgically treated patients difficult.

To identify candidates for surgical treatment, adrenal venous sampling (AVS) is necessary to confirm unilateral disease . However, AVS is a technically demanding procedure, with a mean success rate in non-specialized centres of only 32% . This, and the fact that AVS is not widely available, suggests that a substantial number of patients with unilateral PA are never identified and thereby not considered for surgical treatment .

Rationale, aim and hypotheses

Given the above, medical treatment with MRA has become the de-facto standard treatment for a large number of patients with unilateral PA, despite observational studies indicating that surgical treatment is more effective in terms of improving cardiovascular outcome, quality of life and drug load, and that it is more cost-effective.

In this context the investigators have designed a prospective randomized controlled trial where we aim to compare medical and surgical treatment for unilateral PA. The investigator´s main hypothesis is that surgical treatment (adrenalectomy; standard treatment) results in better QoL at one year of follow-up compared to medical treatment with eplerenone (intervention) in patients with unilateral PA.

The secondary hypotheses are: Surgical treatment is more effective than medical treatment for unilateral PA regarding a) antihypertensive effect, b) improvement in cardiometabolic risk profile, and c) health care consumption (cost-efficiency).

Study Design

The UPA-MEST (Unilateral Primary Aldosteronism - MinEralocorticoid antagonists versusSurgical Treatment) study is an unblinded, prospective, randomized, controlled trial. Eighty patients will be randomized to be either treated surgically with unilateral adrenalectomy or to receive medical treatment with eplerenone. After 12 months of follow-up, medically treated patients will be able to either continue with medical treatment or to be operated with unilateral adrenalectomy.

Participants

80 patients with confirmed unilateral PA, aged 18-70 will participate.

Inclusion and randomization

After unilateral PA has been confirmed, when the patients will be informed about the disease, the patients will be informed orally, and with written information about the study, and asked to participate.

Randomization will be done with random permutated blocks, generated by using a freely available software (www.randomizer.org).

Treatments

Surgical treatment: Minimally invasive surgery is performed via the lateral transperitoneal approach or the posterior retroperitoneal approach, with or without robotic assistance, according to the surgeon's preference. Potassium substitution > 7.5 g will be reduced by 50% on postoperative day (POD) 1, and discontinued on POD 2. Potassium substitution < 7.5 g will be discontinued on POD 1. Preoperative antihypertensive medication will be titrated to a goal blood pressure of 140/90 mmHg (14) or lower. Immunohistochemical method, using monoclonal antibodies identifying the enzymes CYP11B1 and B2, will be used to differentiate between adenoma and hyperplasia.

Medical treatment: The initial dose of eplerenone is 25 mg twice daily. The dose will be increased by 50 mg every fourth week until systolic blood pressure of 140 mmHg and diastolic blood pressure of 90 mmHg or lower has been reached and biochemical control (plasma renin above the middle of the reference range, i.e > ~20 mIU/L) is attained and/or hyperkalemia develops. The maximal dose of eplerenone is 300 mg twice daily. During eplerenone dose titration, the doses of other antihypertensive medications will be reduced or, if possible, discontinued. Also, potassium replacement should be discontinued. In patients who develop significant hyperkalemia (>4.6 mmol/L), the first step is to discontinue ACE inhibitors and/or angiotensin II receptor blocker (ARB). In patients not receiving treatment with ACE inhibitors or ARB, the dose of eplerenone will be decreased by 25-50 mg per day. Similarly, patients on monotherapy with eplerenone who develop very high renin concentrations and/or symptomatic hypotension, the dose of eplerenone should be decreased by 25-50 mg per day. Patients who do not attain optimal blood pressure on the maximal eplerenone dose will continue with other antihypertensive medications. It is expected that creatinine will increase in some patients, reflecting diminished renal hyperfiltration that is characteristic for patients with untreated PA. In these cases, the eplerenone dose should not be automatically reduced, and should only be considered in cases with severely worsening GFR (>1.5 from the baseline value).

Follow-up

Total follow-up time is 24 months. For patients in the MRA arm, there will be a possibility to cross over (opt for surgery) after 12 months. The participants will be followed on at least 7 occasions throughout the study.

Outcome measures

Primary endpoint: The primary endpoint is the difference in improvement of QoL between surgically and medically treated patients at 12 months, measured with EQ5D (total score and the VAS scale).

Secondary endpoints: The secondary endpoints are: 1) Difference in improvement of QoL at 24 months, evaluated with EQ5D, 2) Difference in improvement of QoL at 12 and 24 months, evaluated with the SF-36/RAND-36 questionnaire, 3) The proportion of patients with complete, partial, and absent success of clinical and biochemical outcomes (based on blood pressure, use of antihypertensive drugs, plasma potassium, plasma renin and plasma aldosterone 1) according to the PASO criteria (15) at 12 and 24 months, 4) cardiovascular risk profile at 12 and 24 months, 5) difference in left ventricular mass on echocardiography at 12 and 24 months, 6) difference in renal function, evaluated by measuring eGFR and urinaryalbumin excretion at 12 and 24 months, and 7) total societal cost

Statistics and power calculation

Difference in treatment effects between the two groups will be analysed with paired t-test and Fishers exact test, as well as regression analyses with adjustments for age, gender, duration ofhypertension, as well as blood pressure and number of antihypertensive drugs at baseline.

For power calculation we used quality of life data from Velema et al. (EQ-5D) and Ahmedet al. (RAND SF-36) . With a significance level of 5% and power of 80%, inclusion of 50-54 subjects is needed (25-27 subjects in each treatment arm) to detect a difference betweensurgically and medically treated patients. Allowing for a 20% drop out rate, inclusion is set to 80 subjects (i.e. 40 in each treatment arm).

To ensure external validity, a screening log will be kept at each centre.

Clinical benefits

Contemporary treatment guidelines advocate surgical treatment in patients with unilateral disease. However, since AVS is not always successful, and not widely available, life-long medical treatment is often preferred for patients with PA, without any attempts to find out if they are candidates for curative surgical treatment. It is therefore of great importance to investigate if medical treatment is as effective as surgery in these patients. Currently, a head to head comparison of surgical versus medical treatments for patients with unilateral PA is lacking.

If it turns out that medical treatment is as efficient and safe as surgical treatment for patients with unilateral dominant disease, a large number of patients worldwide will benefit from the study. This concerns patients treated at centres where AVS is not available, patients where the AVS has not been successful as well as patients with unilateral dominant PA who are not considered candidates for surgical intervention. Thus, the study's results have a great potential to be quickly implemented in clinical practice.

Ethical considerations

The main ethical issue to acknowledge is that half of the patients will be randomized to receive medical treatment, i.e. they will not receive surgical treatment that is currently considered to be standard of care for unilateral PA. However, the reasons for considering the trial to be ethical are: a) Medical treatment with mineralocorticoid receptor antagonist forpatients with bilateral PA is effective and safe, b) Thorough information about the study willbe provided before participation, c) Participation is voluntary, d) After 12 months, all medically treated patients will have the option to receive surgical treatment i.e. adrenalectomy.

The study was approved by the Regional Research Ethics Committee in Gothenburg, Sweden on June 3rd, 2020 (DNR 2020-02008).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed unilateral PA
2. Age 18-70 years
3. Candidate for surgical treatment
4. No contraindications for minimally invasive surgery or treatment with MRA
5. Understands oral and written information and provides oral and written informed consent.

Exclusion Criteria:

1. Unwilling or unable to undergo surgery
2. Unwilling to accept medical treatment for 12 months and not receiving standard treatment (surgery)
3. Impaired renal function with eGFR <45 ml/min/1,73m2
4. P-cortisol >138 nmol/L following 1-mg overnight dexamethasone suppression test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2028-05-28 (Estimated); Study Completion 2028-05-28 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) evaluated with EuroQol-5D at 12 months | 1 year
  Improvement in quality of life in surgically and medically treated patients 1 year after treatment of unilateral primary aldosteronism evaluated with EuroQol-5D (EQ-5D-5LTM)
Quality of Life (QoL) evaluated with RAND SF-36 at 12 months | 1 year
  Improvement in quality of life in surgically and medically treated patients 1 year after treatment of unilateral primary aldosteronism evaluated with RAND SF-36.
Quality of Life (QoL) evaluated with EuroQol-5D at 24 months | 2 years
  Improvement in quality of life 2 years after treatment of unilateral primary aldosteronism evaluated with EuroQol-5D (EQ-5D-5LTM)
Quality of Life (QoL) evaluated with RAND SF-36 at 24 months | 2 years
  Improvement in quality of life 2 years after treatment of unilateral primary aldosteronism evaluated with RAND SF-36.

SECONDARY OUTCOMES:
Clinical outcome based on the Primary Aldosteronism Surgical Outcome (PASO) Criteria | 1 year
  To evaluate treatment effects. The proportion of patients with complete, partial or absent clinical success according to the PASO criteria
Biochemical outcome based on the Primary Aldosteronism Surgical Outcome (PASO) Criteria | 1 year
  To evaluate treatment effects. The proportion of patients with complete, partial or absent biochemical success according to the PASO criteria.
Left ventricular mass | 1 year
  To evaluate treatment effects in left ventricular mass by utilizing echocardiography at 12 months
Left ventricular mass | 2 year
  To evaluate treatment effects in left ventricular mass by utilizing echocardiography at 24 months
Glomerular filtration rate (GFR) as a surrogate endpoint of renal function at 12 months | 1 year
  To evaluate changes in renal function by assessment of glomerular filtration rate (GFR)
Albuminuria as a surrogate endpoint of renal function at 24 months | 1 year
  To evaluate changes in renal function by assessment of albuminuria by urine samples (urinary albumin/creatinine ratio)
Total costs | 2 years
  An analysis of total costs for the society will be performed based on patient baseline demographics, an analysis of treatment (in- and outpatient) associated costs, sick leave and disease- and treatment-relatedincome loss to patients and significant others, as well as disease- and treatment-related costs related costs to society.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Ragnarsson, MD, Principal Investigator — Institute of Medicine, Sahlgrenska Academy, University of Gothenburg
Locations (3):
- Sweden (3):
  - University of Gothenburg, Gothenburg
  - Karolinska University Hospital, Stockholm, Sweden., Stockholm
  - Umeå University, Umeå, Sweden., Umeå

IPD SHARING:
Plan to Share IPD: Yes
All data will be available for other researcher upon request
Supporting Information: Study Protocol
Time Frame: The investigators expect to start patient recruitment in February 2023. With an annual AVS rate of 50-70 patients with PA at Gothenburg University Hospital, with an AVS success rate of 97% (13), where approximately 50% are diagnosed with unilateral PA, and a sample size of 80, the estimated accrual time is set to 4 years. To increase the external validity of the study, and to speed up the recruitment period, other centres of excellence for patients with PA will be offered to participate in the study.
Access Criteria: All data will be available for other researcher upon request

REFERENCES:
- [Background] Young WF Jr. Diagnosis and treatment of primary aldosteronism: practical clinical perspectives. J Intern Med. 2019 Feb;285(2):126-148. doi: 10.1111/joim.12831. Epub 2018 Sep 25. PMID 30255616
- [Background] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Background] Monticone S, D'Ascenzo F, Moretti C, Williams TA, Veglio F, Gaita F, Mulatero P. Cardiovascular events and target organ damage in primary aldosteronism compared with essential hypertension: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2018 Jan;6(1):41-50. doi: 10.1016/S2213-8587(17)30319-4. Epub 2017 Nov 9. PMID 29129575
- [Background] Muth A, Ragnarsson O, Johannsson G, Wangberg B. Systematic review of surgery and outcomes in patients with primary aldosteronism. Br J Surg. 2015 Mar;102(4):307-17. doi: 10.1002/bjs.9744. Epub 2015 Jan 20. PMID 25605481
- [Background] Huang WC, Chen YY, Lin YH, Chueh JS. Composite Cardiovascular Outcomes in Patients With Primary Aldosteronism Undergoing Medical Versus Surgical Treatment: A Meta-Analysis. Front Endocrinol (Lausanne). 2021 May 17;12:644260. doi: 10.3389/fendo.2021.644260. eCollection 2021. PMID 34079522
- [Background] Ahmed AH, Gordon RD, Sukor N, Pimenta E, Stowasser M. Quality of life in patients with bilateral primary aldosteronism before and during treatment with spironolactone and/or amiloride, including a comparison with our previously published results in those with unilateral disease treated surgically. J Clin Endocrinol Metab. 2011 Sep;96(9):2904-11. doi: 10.1210/jc.2011-0138. Epub 2011 Jul 21. PMID 21778218
- [Background] Velema M, Dekkers T, Hermus A, Timmers H, Lenders J, Groenewoud H, Schultze Kool L, Langenhuijsen J, Prejbisz A, van der Wilt GJ, Deinum J; SPARTACUS investigators. Quality of Life in Primary Aldosteronism: A Comparative Effectiveness Study of Adrenalectomy and Medical Treatment. J Clin Endocrinol Metab. 2018 Jan 1;103(1):16-24. doi: 10.1210/jc.2017-01442. PMID 29099925
- [Background] Hundemer GL, Curhan GC, Yozamp N, Wang M, Vaidya A. Cardiometabolic outcomes and mortality in medically treated primary aldosteronism: a retrospective cohort study. Lancet Diabetes Endocrinol. 2018 Jan;6(1):51-59. doi: 10.1016/S2213-8587(17)30367-4. Epub 2017 Nov 9. PMID 29129576
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Zhou Y, Wang D, Jiang L, Ran F, Chen S, Zhou P, Wang P. Diagnostic accuracy of adrenal imaging for subtype diagnosis in primary aldosteronism: systematic review and meta-analysis. BMJ Open. 2020 Dec 31;10(12):e038489. doi: 10.1136/bmjopen-2020-038489. PMID 33384386
- [Background] Schirpenbach C, Segmiller F, Diederich S, Hahner S, Lorenz R, Rump LC, Seufert J, Quinkler M, Bidlingmaier M, Beuschlein F, Endres S, Reincke M. The diagnosis and treatment of primary hyperaldosteronism in Germany: results on 555 patients from the German Conn Registry. Dtsch Arztebl Int. 2009 May;106(18):305-11. doi: 10.3238/arztebl.2009.0305. Epub 2009 May 1. PMID 19547646